CLINICAL TRIAL: NCT01275508
Title: Prospective, Monocentric, Open-label, Clinical Phase 1 Study to Demonstrate the Safety and Tolerability of FITC-Adalimumab After Single Topical Administration to the Intestinal Mucosa During Endomicroscopy in Patients With Crohn's Disease
Brief Title: Safety and Tolerability of FITC-Adalimumab Administration During Confocal Laser Endomicroscopy of the Gut
Acronym: FA-Crohn
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FITC-ADA 01-2010; 2010-018959-99 (EudraCT Number)
Record Dates: First submitted 2011-01-07; First posted 2011-01-12 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Crohn's Disease
Keywords: Subjects with active Crohn's disease; Safety and tolerability of FITC-Adalimumab; Intestinal topical application
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FITC-Adalimumab (Experimental)
  Interventions: Drug: FITC-Adalimumab

INTERVENTIONS:
Drug: FITC-Adalimumab — The study product FITC-Adalimumab will be topically applied via a spray catheter to the intestinal mucosa of Crohn's disease patients during endomicroscopy of the gut. One mL of the diluted study product will be applied each time to overall four selected intestinal areas at a concentration of 20 μg/mL respectively (equivalent to 20 μg of FITC-Adalimumab per area). Total amount applied will be 80 μg FITC-Adalimumab per patient.

SUMMARY:
The scientific objective of the project is to evaluate if the topical administration of Fluoresceinisothiocyanate (FITC)-Adalimumab during the endomicroscopic examination of the gut in Crohn's disease (CD) patients shows an acceptable safety profile. Another objective is to explore whether the use of FITC-Adalimumab as a predictive biomarker might reliably predict patient response to Adalimumab therapy and hence enable optimized utilization of this treatment option.

ELIGIBILITY:
Inclusion Criteria:

Trial subjects must meet all of the following inclusion criteria:

* Male and female subjects from 18 to 70 years of age who are capable of giving informed consent without any restrictions
* Endoscopically and histologically confirmed diagnosis of Crohn's disease (CD)
* Manifestation of CD in the colon and/or in the terminal ileum
* Currently active CD with a CDAI score >150
* Clinically inadequate response of CD to systemic glucocorticoids and/or immunosuppressants (azathioprine, 6-mercaptopurine, methotrexate) or glucocorticoid-dependent CD or any contraindication to glucocorticoids
* Indication for treatment with Adalimumab
* Indication for intestinal confocal laser endomicroscopy prior to institution of adalimumab therapy
* Subject is mentally capable of understanding the nature and purpose/conduct of the clinical trial and of following the study staff's instructions
* Subject has given written informed consent after being informed by an investigator

Female subjects additionally must meet at least one of the following criteria:

* Must be menopausal (at least 12 months' natural amenorrhea or 6 months' amenorrhea with serum FSH >40 mU/mL) or
* Must have undergone bilateral oophorectomy or hysterectomy or
* Must be a regular, correct, and reliable user of a contraceptive method with a failure rate of <1% per year (such as oral contraceptives, implants, depot shots, intrauterine device, hormone coil)
* Must have a vasectomized partner

Exclusion Criteria:

* Subjects must not meet any of the following exclusion criteria:
* Impaired blood clotting (prothrombin rate <50% and/or PTT >55 sec and/or a platelet count of <50,000/μL)
* Pregnancy and lactation

Contraindications to treatment with adalimumab:

* Moderate to severe heart failure (NYHA Class III/IV)
* Active tuberculosis
* Severe acute infections, e.g. sepsis
* Opportunistic infections including invasive fungal infections

  * Known hypersensitivity to any of the ingredients of the study product or to any drug with a similar chemical structure
  * Treatment with beta-receptor blocking agents (because of altered symptoms in case of possible anaphylactic reactions to IV fluorescein)
  * Any other condition or medical treatment that, in the investigator's judgment, is not compatible with participation in the trial
  * Individuals who are in a relationship of dependence on or employed by the sponsor or any of the investigators
  * Planned prolonged stay outside the region of the study site, preventing the subject from returning for scheduled visits
  * Participation in any other clinical trial or administration of any investigational drug within the last four weeks prior to the screening visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Fluoresceinisothiocyanate (FITC)-Adalimumab | 3 months
  Local Tolerability:
  All intestinal mucosal adverse events observed following administration of FITC-Adalimumab.
  Systemic Safety and Tolerability:
  Number of SARs during the observation period, i.e., number of SAEs whose occurrence is due to the use of FITC-Adalimumab in this clinical trial.
  Number of SAEs during the observation period. Number of AEs during the observation period.

SECONDARY OUTCOMES:
Visual identification of FITC-Adalimumab positive intestinal mucosal cells | One minute after administration of FITC-Adalimumab
  Visual identification (yes/no) of FITC-Adalimumab positive intestinal mucosal cells by confocal laser endomicroscopy following labeling with FITC-Adalimumab
Number of FITC-Adalimumab positive intestinal mucosal cells | One minute after administration of FITC-Adalimumab
  Number of FITC-Adalimumab positive intestinal mucosal cells as identified by confocal laser endomicroscopy following labeling with FITC-Adalimumab
Correlation between the number of FITC-Adalimumab positive intestinal mucosal cells in inflamed gut sections and therapeutic response to Adalimumab therapy. | Three months after administration of FITC-Adalimumab
  Correlation between the number of FITC-Adalimumab positive intestinal mucosal cells in inflamed gut sections and therapeutic response.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Neurath, MD PhD, Study Director — Medizinische Klinik I, University Hospital Erlangen; Raja Atreya, MD, PhD, Principal Investigator — Medizinische Klinik I, University Hospital Erlangen
Locations (1):
- Medizinische Klinik I, University Hospital Erlangen, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Colombel JF, Sandborn WJ, Rutgeerts P, Enns R, Hanauer SB, Panaccione R, Schreiber S, Byczkowski D, Li J, Kent JD, Pollack PF. Adalimumab for maintenance of clinical response and remission in patients with Crohn's disease: the CHARM trial. Gastroenterology. 2007 Jan;132(1):52-65. doi: 10.1053/j.gastro.2006.11.041. Epub 2006 Nov 29. PMID 17241859
- [Background] Keller R, Winde G, Terpe HJ, Foerster EC, Domschke W. Fluorescence endoscopy using a fluorescein-labeled monoclonal antibody against carcinoembryonic antigen in patients with colorectal carcinoma and adenoma. Endoscopy. 2002 Oct;34(10):801-7. doi: 10.1055/s-2002-34254. PMID 12244502
- [Background] Kiesslich R, Burg J, Vieth M, Gnaendiger J, Enders M, Delaney P, Polglase A, McLaren W, Janell D, Thomas S, Nafe B, Galle PR, Neurath MF. Confocal laser endoscopy for diagnosing intraepithelial neoplasias and colorectal cancer in vivo. Gastroenterology. 2004 Sep;127(3):706-13. doi: 10.1053/j.gastro.2004.06.050. PMID 15362025
- [Background] Kiesslich R, Goetz M, Vieth M, Galle PR, Neurath MF. Technology insight: confocal laser endoscopy for in vivo diagnosis of colorectal cancer. Nat Clin Pract Oncol. 2007 Aug;4(8):480-90. doi: 10.1038/ncponc0881. PMID 17657253